CLINICAL TRIAL: NCT06415240
Title: Assistant Clinical Nurse Manager Working in Neonatal Intensive Care Unit
Brief Title: Effect of Facilitated Tucking and Gentle Human Touch on Procedural Pain Among Neonates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Nazma Hamid, Assistant Clinical Nurse Manager, Shifa International Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STMU
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Non Pharmacological Pain Management
Keywords: Non Pharmacological Pain Management; Neonates; Procedural Pain
MeSH Terms: conditions — Pain, Procedural | interventions — Facilitated Tucking

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant, Investigator
Masking Description: As participants are neonates, they are not able to judge any intervention. Data is being collected by an independent data collector and pain scoring is also planned to be done by an independent Research Assistant. So, an investigator is masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facilitated Tucking (Experimental): A non pharmacological intervention to be implemented during arterial prick.
  Interventions: Other: Facilitated Tucking
- Gentle Human Touch (Experimental): A non pharmacological intervention to be implemented during arterial prick.
  Interventions: Other: Gentle Human Touch
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Other: Facilitated Tucking — Facilitated Tucking is a position to be adopted for pain relief in neonates.
  Arms: Facilitated Tucking
Other: Gentle Human Touch — while gentle human touch is caressing on head for pain relief.
  Arms: Gentle Human Touch

SUMMARY:
This is a Randomized Control Trial intended to investigate the effect of two non-pharmacological interventions on procedural pain among neonates.

DETAILED DESCRIPTION:
The Study Design is a Randomized Control Trial, intended to investigate the effect of facilitated tucking and gentle human touch on procedural pain among neonates (age 28 days). Neonatal Infant Pain Scale will be used for pain scoring, data will be collected by recording demographic variables for all neonates and then capturing a video recording for pain scoring by an independent research assistant.

ELIGIBILITY:
Inclusion Criteria:

1. Both term and preterm neonates.
2. APGAR scores of a minimum of 6 at one minute and 8 at 5 minutes
3. Admitted to the Neonatal Intensive Care Unit
4. Undergoing arterial prick for the first time.

Exclusion Criteria:

1. Documented birth asphyxia
2. Congenital anomalies
3. Neurological diagnosis,
4. ventilated with paralysis
5. Extremely premature newborns (Gestational age < 28 weeks)

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale | Before,During Arterial Prick and after three minutes
  scoring of pain based on a scale used in neonates both for term and pre term babies.( Minimum Pain Score 0, Maximum 7, Higher number indicates the worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nazma Hamid, MSN, Principal Investigator — Shifa Tameer E Millat Univesrity
Locations (2):
- Pakistan (2):
  - Pakistan Institute of Medical Sciences, Islamabad
  - Shifa Tameer E Millat University, Islamabad

IPD SHARING:
Plan to Share IPD: No
Not intended